CLINICAL TRIAL: NCT01562600
Title: Nexium Capsules Specific Clinical Experience Investigation for Long-term Use Concerning Prevention of Recurrence of Gastric Ulcer or Duodenal Ulcer With NSAIDs
Brief Title: Nexium Capsules Non-steroidal Anti-inflammatory Drug (NSAID) Specific Clinical Experience Investigation
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D961HC00012
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Gastric Ulcer; Duodenal Ulcer
Keywords: NSAIDs; Gastric ulcer or duodenal ulcer; Nexium
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Nexium

SUMMARY:
The purpose of this investigation is to collect following data in patients given Nexium capsule (Nexium) for long term in usual-post-marketing therapy to prevention of recurrence of gastric ulcer or duodenal ulcer with non-steroidal anti-inflammatory drug (NSAID).

DETAILED DESCRIPTION:
Nexium capsules Specific Clinical Experience Investigation for long-term use concerning prevention of recurrence of gastric ulcer or duodenal ulcer with NSAIDs

ELIGIBILITY:
Inclusion Criteria:

-Patients who are given NSAIDs for long terms to control pain due to disease such as rheumatoid arthritis and osteoarthritis, and given Nexium to suppress recurrence of gastric ulcer or duodenal ulcer.

Exclusion Criteria:

* Patients having gastric ulcer/duodenal ulcer when Nexium is started (Active phase (A1, A2) or healing phase (H1, H2) of Sakita-Miwa classification on endoscopy)
* Patients who had been given Nexium for suppression of recurrence of gastric ulcer/duodenal ulcer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are given NSAIDs for long terms to control pain due to disease such as rheumatoid arthritis and osteoarthritis, and given Nexium to suppress recurrence of gastric ulcer or duodenal ulcer.
  (Patients who have previous experience of Nexium given in the treatment for gastric ulcer or duodenal ulcer can be registered to this S-CEI.)
Sampling Method: Non-Probability Sample
Enrollment: 1634 (Actual)
Dates: Start 2012-04-19 (Actual); Primary Completion 2015-08-27 (Actual); Study Completion 2015-08-27 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Drug Reactions | 1 Year
  Adverse event incidence

SECONDARY OUTCOMES:
Non-recurrence rate of peptic ulcer | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Yoshida, MD, Study Director — AstraZeneca
Locations (46):
- Japan (46):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

REFERENCES:
- See also: AZ_Synopsis_D961HC00012_STUDY_REPORT_SUMMARY_revised — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=707&filename=AZ_Synopsis_D961HC00012_STUDY_REPORT_SUMMARY_revised.pdf
- See also: K. Sakamoto, M. Nii, T. Tokimoto and Y. Takumi Esomeprazole (Nexium) Specific Clinical Experience Investigation for Long-term Use in the Prevention of the Recurrence of Gastric or Duodenal Ulcer with NSAIDs Jpn Pharmacol Ther, 47(7), 1043 - 1057, 2019 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D961HC00012&attachmentIdentifier=8bc7ac27-ffcc-42ee-9237-a5b2c2efb304&fileName=Nexium_SCEI_NSAID_LongTerm_Protocol_ver2_redacted.pdf&versionIdentifier=